CLINICAL TRIAL: NCT05652634
Title: Chronic Stress as a Risk Factor for Long COVID
Acronym: StressLoC
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: University of Klagenfurt (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Christian Fazekas, Senior Scientist at Clinical Division of Medical Psychology, Psychosomatics and Psychotherapy, Principal Investigator, Medical University of Graz
Other Study IDs: KLI 1100-B
Record Dates: First submitted 2022-12-14; First posted 2022-12-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Long COVID; Acute COVID-19
Keywords: Chronic stress; Long COVID; Mental health; Cognitive function; Stress-related biomarkers
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Proinflammatory cytokines
  2. metabolites of the kynurenine pathway
  3. catecholamines
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The disease caused by the pathogen SARS-CoV-2 is known as coronavirus disease with the acronym COVID-19. The acute phase of this condition typically lasts one to two weeks and usually results in a full recovery. However, in about 10-30% of those affected, the symptoms persist for more than four weeks after the onset of the disease. In this case, there is an ongoing COVID-19 illness known as long COVID. Long COVID can persist for many months and cause significant distress and limitations to those affected due to the long-term health consequences.

The causes of long COVID are still unclear and, accordingly, therapeutic measures are still insufficiently developed. It is assumed that long COVID can in principle affect anyone. Age, gender, obesity and the number of symptoms during an acute COVID-19 illness are discussed as risk factors for long COVID. Another potential risk factor for developing long COVID could be chronic stress, which has been shown to put a strain on the immune system. It is known from infections with other coronaviruses and other viral respiratory diseases that chronic stress can lead to prolonged illness and limited recovery. The aim of this study is to systematically examine chronic stress, as it existed before infection with the coronavirus, as a possible risk factor for long COVID.

For this purpose, 600 people who have been proven to be infected with SARS-CoV-2 and have developed symptoms of COVID-19 will be included in this study.

DETAILED DESCRIPTION:
Wider research context / theoretical framework: The pathophysiology leading to symptom persistence after acute COVID-19, defining long COVID, is widely unknown. Chronic stress may be a risk factor for long COVID as it can impair immune regulation and induce exaggerated inflammatory responses. It is known to negatively influence upper respiratory infections and was found to be associated with long-term symptoms following other coronavirus infections (SARS). In addition, chronic stress is an established risk factor for unspecific functional symptoms and mental health impairment. Data on these issues are scanty, however much-needed for developing proper interventions.

Hypotheses/research questions/objectives: The primary aim of the study is to analyze the influence of chronic stress on symptom persistence in COVID-19. The study team hypothesizes that elevated levels of pre-existing self-reported chronic stress measured at the beginning of infection predict a higher proportion of patients with symptom persistence at one month after testing positive for SARS-CoV-2 infection (primary outcome). Secondary aims are to investigate the influence of chronic stress on medium- to long-term mental health outcome. In addition, the researchers longitudinally investigate chronic stress, stress-related biomarkers and allostatic load in patients with symptom persistence as compared to recovered patients.

Approach/methods: This is a longitudinal prospective observational study designed according to STROBE guidelines in persons newly tested positive for SARS-CoV-2 infection by qPCR with symptoms of acute COVID-19. Monitoring of COVID-19-related symptoms and symptom persistence is conducted online, by phone and in outpatient clinic visits. Pre-existing chronic stress is investigated by questionnaires on perceived stress and negative life events and by analysis of hair cortisol concentrations prior to infection. Collection of blood allows measurement of SARS-CoV-2 antibodies, stress-related biomarkers and the calculation of allostatic load. Baseline and longitudinal data collection encompasses comorbidities, regular medication, screening for anxiety, depression, acute stress symptoms, and cognitive function.

Level of originality/innovation: This is the first study prospectively investigating chronic stress as a risk factor for long COVID and associated mental health impairment by a multimodal approach. In addition, the researchers probe for stress-related biomarkers associated with symptom persistence and also investigate the impact of protective factors, such as resilience, psychosomatic competence and social support, on symptom persistence. Two novel bio-psycho-social assessment tools contribute to the results of this study. Results of this project will lead to innovative preventive and treatment interventions targeting symptom persistence and mental health sequelae after acute COVID-19.

Primary researchers: Christian Fazekas (PI), Nandu Goswami, Barbara Hanfstingl, Voyko Kavcic.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years); qPCR-test positive for SARS-CoV-2 infection; symptom(s) of acute COVID-19; inclusion within defined timeframe of one week after testing; data collection online, by phone and at study visits feasible

Exclusion Criteria:

* Insufficient knowledge of German language; lengths of hair at rear vertex less than 2 cm; pregnancy or postpartum less than 3 months; refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After having been tested positive for SARS-CoV-2 and having received the invitation to participate in this study by the local health authority of the City of Graz, or the health authority of the Province of Styria, persons interested can visit the study website and sign in for getting contacted by the study team.
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Symptom persistence beyond four weeks from the onset of acute symptoms of COVID-19 (subacute/ongoing symptomatic COVID-19). | Symptom persistence at one month after having tested positive for SARS-CoV-2 infection (subacute/ongoing symptomatic COVID-19)
  Application of the Long COVID Symptom Tool and Impact Tool (LC-ST and LC-IT)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Division of Medical Psychology, Psychosomatics and Psychotherapy, Graz, Styria, Austria